CLINICAL TRIAL: NCT01265836
Title: Dyslipidemia Treatment in Thailand and Cardiovascular Outcomes
Acronym: DEMAND
Status: Withdrawn | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Marketing Company Medical Director, AstraZeneca
Other Study IDs: NIS-CTH-DUM-2010/1
Record Dates: First submitted 2010-12-14; First posted 2010-12-23 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia Treatment and Cardiovascular Outcomes
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to establish the proportion of patients on lipid-lowering pharmacological treatment (statin or combination) reaching the LDL-C goals according to the updated 2004 National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) guidelines.

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent, Female or male aged = 18 years
* Patients eligible for treatment of dyslipidemia with statins, according to the current guidelines NCEP ATPIII about Dyslipidemias and Atherosclerosis Prevention Receiving lipid-lowering drug treatment for at least 15 days.

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to either AstraZeneca staff or staff at the study site).
* Previous enrolment or randomisation of treatment in the present study
* Participation in a clinical study during the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Provision of subject informed consent
  2. Female or male aged = 18 years
  3. Patients eligible for treatment of dyslipidemia with statins, according to the current guidelines NCEP ATPIII about Dyslipidemias and Atherosclerosis Prevention.
  4. Receiving lipid-lowering drug treatment for at least 15 days.
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
The number (#) of subjects achieving the LDL-C goals according to updated 2004 NCEP ATP III guidelines. | 1 year
The percent (%) of subjects achieving the LDL-C goals according to updated 2004 NCEP ATP III guidelines. | 1 year

SECONDARY OUTCOMES:
The number of subjects achieving the LDL-C goals according to the updated 2004 NCEP ATP III guidelines for several subject subsets | 1 year
The number of the secondary event rate of cerebrovascular patients on lipid-lowering pharmacological treatment (statin or combination) who reaching and non-reaching the LDL-C goals according to the updated 2004 NCEP ATP III guidelines for 1 | 1 year
The number of the secondary event rate cardiovascular patients on lipid-lowering pharmacological treatment (statin or combination) who reaching and non-reaching the LDL-C goals according to the updated 2004 NCEP ATP III guidelines for 1 year | 1 year
The percentage of subjects achieving the LDL-C goals according to the updated 2004 NCEP ATP III guidelines for several subject subsets | 1 year
The percent of the secondary event rate of cerebrovascular patients on lipid-lowering pharmacological treatment (statin or combination) who reaching and non-reaching the LDL-C goals according to the updated 2004 NCEP ATP III guidelines for 1 | 1 year
The percent of the secondary event rate cardiovascular patients on lipid-lowering pharmacological treatment (statin or combination) who reaching and non-reaching the LDL-C goals according to the updated 2004 NCEP ATP III guidelines for 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Apichard Sukonthasarn, Prof.M.D., Principal Investigator — Maharaj Nakorn Chiangmai Hospital Cardiovascular division, Department of Internal Medicine, Faculty of Medicine, Chiangmai University